CLINICAL TRIAL: NCT03439696
Title: Needlescopic-assisted Uniportal VATS Versus Conventional Uniportal VATS. A Randomized Prospective Noninferiority Study
Brief Title: Needlescopic-assisted Uniportal vs Uniportal VATS
Acronym: UNeed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRB of NTUH Hsin-Chu Branch (Other)
Responsible Party: Sponsor-Investigator, IRB of NTUH Hsin-Chu Branch, National Taiwan University Hospital Hsin-Chu Branch, National Taiwan University Hospital Hsin-Chu Branch
Organization: National Taiwan University Hospital Hsin-Chu Branch (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106-067-F
Record Dates: First submitted 2018-02-07; First posted 2018-02-20 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer; Lung Cancer Metastatic; Bullous Disease Lung; Nodule Solitary Pulmonary; Mediastinal Tumor
Keywords: Thoracoscopy; VATS; Needlescopy; Uniportal
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule; Mediastinal Neoplasms | interventions — Thoracoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needlescopic-assisted (Experimental): Thoracoscopic surgery performed with the fashion of single 2.5-3.5 cm intercostal incision and 1-2 additional 2-3 mmm needlescopic ports.
  Interventions: Procedure: Thoracoscopic surgery
- Uniportal (Active Comparator): Conventional uniportal VATS with single 2.5-3.5 cm intercostal incision
  Interventions: Procedure: Thoracoscopic surgery

INTERVENTIONS:
Procedure: Thoracoscopic surgery — Video-assisted thoracoscopic surgery for pulmonary or mediastinal lesions.

SUMMARY:
The investigators' study aims is to evaluate the safety and efficacy of uniportal VATS under assistance of needlescopic instruments through additional 2-3 mm ports compared to conventional uniportal VATS in patients with lung lesions.

ELIGIBILITY:
Inclusion Criteria:

Lung or mediastinal disease requiring thoracoscopic surgery

Exclusion Criteria:

Thoracoscopic esophagectomy Decortication for empyema

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Pain scale POD 3 | 3 days
  Post-operative day 3 pain scale documented using Visual Analogue Scale (VAS)
Pain scale POD 5 | 5 days
  Post-operative day 5 pain scale documented using Visual Analogue Scale (VAS)
Hospital stay | 14 days
  Post-operative hospital stay
Post-operative 3 month neuralgia | 3 months
  Out patient documented using PainDETECT questionnaire (PD-Q)
Post-operative 6 month neuralgia | 6 months
  Out patient documented using PainDETECT questionnaire (PD-Q)

SECONDARY OUTCOMES:
Cost | 14 days
  Total hospital cost
Surgical time | 1 day
  Time spend in surgery
Surgical bleeding | 1 day
  Blood loss during operation
Opioid using dosage | 14 days
  Total opioid equivalent dose used during post-operative course

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-kuei Nien, Principal Investigator — National Taiwan University Hospital Hsinchu Branch
Locations (1):
- National Taiwan University Hospital, Hsin-Chu Branch, Taipei, Hsin-Chu County, Taiwan